CLINICAL TRIAL: NCT07201792
Title: Effects of Early Physiotherapy Program on the Infants in the Neonatal Intensive Care Unit: A Randomized Controlled Clinical Trial
Brief Title: Effects of Early Physiotherapy Program on the Infants in NICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Hatice Adiguzel, Associate Profesor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACUT PT IN NICU
Record Dates: First submitted 2025-09-15; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Infants Admitted to Neonatal Units; NICU; NICU Infants; Family Centered Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early physiotherapy (Experimental): A physiotherapy program tailored to the needs of infants from families who volunteer will be implemented until and including discharge. Parents of all infants discharged from the NICU will receive advice on holding, carrying, and positioning.
  Interventions: Other: Early Physiotherapy
- Standard of care (No Intervention): Infants from families who cannot attend physiotherapy for any reason (those living outside the province, those who cannot attend treatment sessions at the same frequency, working parents) will constitute the control group if they can come to the evaluations.

INTERVENTIONS:
Other: Early Physiotherapy — The early physiotherapy program will begin when the infant is stable and continue until discharge. Depending on the infant's gestational age and respiratory needs, chest physiotherapy, developmental physiotherapy, or both will be administered, if necessary. The early family collaborative physiotherapy program will begin from the first day the infant is stable and parental contact is established, and will consist of routine-based care and family education programs that include therapeutic holding, carrying, positioning, and sucking facilitation to stimulate postural responses. The physiotherapy group will receive a routine-based family collaborative early intervention program. This program will be based on a model of goal-oriented active motor learning and sensory strategy development in an enriched environment, and will include family education programs that integrate holding, carrying, and positioning training into daily routines. All parents will participate in the training.
  Arms: early physiotherapy

SUMMARY:
High-risk of Infants are defined as one with a history of negative environmental and biological factors that could lead to neuromotor developmental problems. This heterogeneous group encompasses premature babies born at less than 37 weeks, term babies with low birth weight (LBW), or babies with developmental delays due to various causes.Studies have highlighted that individual developmental care, family education, kangaroo care, and early physiotherapy approaches applied to at-risk infants in the neonatal intensive care unit (NICU) enhance infant development. However, further research is needed to determine the most effective interventions for infants who are more environmentally at risk and biologically vulnerable. Studies investigating the effectiveness of early intervention methods initiated in the NICU on the motor, cognitive, and behavioral outcomes of premature infants have highlighted that postural control interventions or physiotherapy consisting of developmental care programs implemented in the neonatal period improve motor development in the short term, but parent-implemented motor interventions are more effective in improving infants' cognitive and motor outcomes in the long term.The aim of this study is to examine the effects of family-based early physiotherapy approaches applied to at-risk infants in the NICU on motor, cognitive, language development and developmental outcomes at term age and in the long term (adjusted 3, 6, 9, 12 months).

ELIGIBILITY:
Inclusion Criteria:

* Newborns diagnosed with periventricular hemorrhage (PVH), intracranial hemorrhage (ICH), cystic PVL, HIE, kernicterus, perinatal asphyxia, neonatal sepsis, necrotizing enterocolitis (NEC), retinopathy of prematurity (ROP), RDS, or BPD.
* Newborns receiving oxygen or mechanical ventilation (MV) support.
* Infants with a 5-minute Apgar score <3, <37 weeks' gestation, <1500 g preterm, or prematurity due to multiple births.

Exclusion Criteria:

* Newborns with congenital malformations (spina bifida, congenital muscular torticollis, arthrogryposis multiplex congenita, etc.), babies diagnosed with metabolic and genetic diseases (down syndrome, spinal muscular atrophy, duchenne muscular dystrophy, etc.)

Ages: 28 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Prechtl's General Movements (GMs) Assessment | writhing movement betweeen birth and 8 weeks of age, Fidgety movements between 12 and 20 weeks of age
  Prechtl's General Movements (GMs) Assessment: General movements (GMs) are the spontaneous movement repertoire present from early fetal life until the 20th week postpartum. They are "writhing" until the 8th week postpartum and then "fidgety" until approximately the 20th week. Heinz Prechtl demonstrated the validity and reliability of this method by determining that infants without fidgety movements between 3 and 5 months of age are at high risk of developing CP. Video recordings will begin in the NICU 3 days after birth during the preterm period. All infants will be examined for writhing and fidgety movements (FM) using the video recordings. Movements during the preterm and writhing periods will be classified as PR, CS, and Ch GMs or normal. Movements during the fidgety period will be recorded as F+ or F++ when normal, AF when abnormal, or F- when not observed. Motor optimality scores will also be calculated for all infants during the fidgety period.
Hammersmith Infant Neurological Examination (HINE) | It will be applied at the adjusted 2nd, 3rd, 6th, 9th and 12th months.
  The HINE is a simple, standardized, and scoreable test for the clinical neurological assessment of infants aged 2-24 months. It consists of three sections: (1) a neurological examination that assesses cranial nerve function, posture, movements, tone, reflexes, and reactions; (2) motor milestones; and (3) behavior. Each of the 26 items on the test is first scored individually (0, 1, 2, 3, or half-point). A total score is then calculated, with a maximum score of 78. The total score is classified as optimal or suboptimal. Optimal scores are based on the frequency distribution of neurological findings in the population observed in at least 90% of infants in the age range studied. Higher scores indicate better neurological status.
BAYLEY-III Infant and Child Development Assessment Scale (BAYLEY-III) | at 3, 6 and 12th months
  The BSID-III is a neurocognitive assessment used to monitor the development of infants aged 0-42 months. It has five domains: cognitive, language, motor, social-emotional, and adaptive functions. This study will assess only the first three domains. Cognitive, language, and fine and gross motor skills will be assessed. A composite score is calculated for each domain (mean 100±15). A composite score below 2 standard deviations (SD) (<70) is considered a severe delay across all domains.

SECONDARY OUTCOMES:
Sociodemographic form | first day of the assessment
  Prenatal/perinatal risks (MRI, cUS results, diagnosis, neurological evaluation) of all infants and their parents will be obtained from hospital records after treatment.
Hammersmith Neonatal Neurological Examination | 3 days after birth and corrected postterm 40±2 weeks
  The examination developed by Dubowitz standardized optimality scores by evaluating low-risk term and high-risk preterm infants at term age. The scale consists of a 34-item proforma. This proforma includes tone (10), tone patterns (5), reflexes (6), movements (3), abnormal signs (3), and behavior (7). All items are scored from 1 to 3 (half points are also possible). Higher scores indicate better neurological status.
Body Mass Index (BMI) | baseline
  Birth weight in kilograms, height in meters will be recorded. Weight and height will be combined to report BMI in kg/m2.

CONTACTS AND LOCATIONS:
Overall Officials: hatice adıgüzel tat, Associate Professor, Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (1):
- Kahramanmaraş Sütçü imam University, Kahramanmaraş, Onikişubet, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No